CLINICAL TRIAL: NCT01036360
Title: Regulation of the Energy Balance Following an Acute Exercise in Metabolic Chambers: Effect of the Exercise Intensity, Age and Weight Status
Brief Title: Acute Exercise and Energy Balance Regulation: Effect of Intensity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Regional Program for Clinical Research 2009 (PHRC 2009) (Unknown); Thermal Institution of Brides les Bains (FRANCE) (Unknown)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Other Study IDs: CHU-0063
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Obesity
Keywords: Obesity; Acute exercise; Intensity of exercise; Energy balance regulation; Appetite
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Defined population

GROUPS / COHORTS (1):
- physical activity
  Interventions: Other: metabolic chamber

INTERVENTIONS:
Other: metabolic chamber — 20 adolescent boys (10 obese and 10 leans) and 20 men (10 obese and 10 lean) will complete a sub-maximal test on a ergo cycle to draw their linear relationship between VO2 and Fc. Then they will enter a metabolic chamber three times, for 24 hours each

SUMMARY:
Physical activity is mainly considered and use for its impact on energy expenditure in the treatment of obesity, and less is known concerning its indirect effects on energy intake. The aim of this work is to clarify the impact of an acute bout of exercise, depending on its intensity (high versus low), on the following energy intake and nutrient utilization, in obese and non-obese boys and men.

DETAILED DESCRIPTION:
20 adolescent boys (10 obese and 10 leans) and 20 men (10 obese and 10 lean) will complete a sub-maximal test on a ergo cycle to draw their linear relationship between VO2 and Fc. Then they will enter a metabolic chamber three times, for 24 hours each. A first session will be considered as sedentary, and volunteers will remain inactive. During the second and third session, they will have to complete a cycling test generating an energy expenditure of 400 Kcal, once at low intensity (40%VO2max) and once at high intensity (70% VO2max). Those three sessions will be realized in a randomized order with an interval of at least 7 days and urinary collection over the 24hours will be done during all the sessions. At the beginning of the protocol, blood samples will be taken, body composition assessed by DXA and adiposity location evaluated by MNR.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Adults between 18 to 30 years old and adolescents between 12 and 15 years old
* Body mass index :

  * lean adults : 20 <BMI< 25 kg.m²
  * obese adults : 30<BMI<38 kg.m²
  * lean adolescents: BMI <90th percentile
  * obese adolescents: BMI>97th percentile
* Affiliated to National Health Insurance
* Subject giving his written informed consent
* Subject considered as normal after clinical examination and medical questionnaire.

Exclusion Criteria:

* Chronic pathologies : cardiovascular diseases, cancer, chronic inflammation diseases, renal, intestinal impairments
* Refusal to be registered on the National Volunteers Data file
* Being in exclusion on the National Volunteers Data file
* Practising intensive physical exercise
* Heavy consumer of alcohol or/and tobacco
* Previous medical and/or surgery judged by the investigator as incompatible with this study

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 adolescent boys (10 obese and 10 leans) and 20 men (10 obese and 10 lean
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The amount of energy intake over the 24 hours is the primary outcome. It will be assessed during the 3 experimental conditions: sedentary, low intensive exercise, high intensive exercise | over the 24 hours

SECONDARY OUTCOMES:
Appetite feeling and substrate utilization are the two second outcomes. It will be assessed during the 3 experimental conditions: sedentary, low intensive exercise, high intensive exercise | with an interval of at least 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Corinne BOUTELOUP, Principal Investigator — CHU Clermont-Ferrand (CRNH)
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Aucouturier J, Thivel D, Isacco L, Fellmann N, Chardigny JM, Duclos M, Duche P. Combined food intake and exercise unmask different hormonal responses in lean and obese children. Appl Physiol Nutr Metab. 2013 Jun;38(6):638-43. doi: 10.1139/apnm-2012-0246. Epub 2013 Jan 10. PMID 23724881
- [Derived] Thivel D, Isacco L, Montaurier C, Boirie Y, Duche P, Morio B. The 24-h energy intake of obese adolescents is spontaneously reduced after intensive exercise: a randomized controlled trial in calorimetric chambers. PLoS One. 2012;7(1):e29840. doi: 10.1371/journal.pone.0029840. Epub 2012 Jan 17. PMID 22272251
- [Derived] Thivel D, Isacco L, Taillardat M, Rousset S, Boirie Y, Morio B, Duche P. Gender effect on exercise-induced energy intake modification among obese adolescents. Appetite. 2011 Jun;56(3):658-61. doi: 10.1016/j.appet.2011.02.020. Epub 2011 Mar 2. PMID 21376093